CLINICAL TRIAL: NCT02797353
Title: Strengthening Maternal Neonatal and Child Health Services in a Rural District of Pakistan
Acronym: SRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: The International Federation of Red Cross and Red Crescent Societies (Other)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Associate Professor, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2787-Ped-ERC-13
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Antepartum Hemorrhage; Postpartum Hemorrhage; Anemia; Eclampsia; Neonatal Sepsis; Birth Asphyxia; Diarrhoea; Pneumonia
MeSH Terms: conditions — Postpartum Hemorrhage; Anemia; Eclampsia; Neonatal Sepsis; Asphyxia Neonatorum; Diarrhea; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Experimental): Antenatal Care, Post natal care, Skilled birth attendance, recognition and referrals of complicated cases, immunization
  Interventions: Other: Maternal Neonatal and Child Health Interventions
- Control (No Intervention): This arm will receive the standard MNCH services as outlined in the MNCH policy of Government of Pakistan

INTERVENTIONS:
Other: Maternal Neonatal and Child Health Interventions — Antenatal care, postnatal care, skilled birth attendance, recognition and referral of complicated cases, immunization
  Arms: Intervention Arm

SUMMARY:
The Maternal Neonatal and Child health indicators in District Dadu of Pakistan portrays a dismal pictures and after the floods of 2010-2011 the health infrastructure of this district was badly affected. Aga Khan University Pakistan is intending to implement a service delivery project for the improvement of Maternal Neonatal and Child health situation through evidence based MNCH interventions.

DETAILED DESCRIPTION:
The Aga Khan University is implementing together with its local partners a MNCH project in five Union Councils (UC) in Dadu District in Sindh Province. The project will scale up the already existing health services for MNCH in the district referral hospital and the five Basic Health Units (BHUs), one in each UC. Institutional based services as well as their scope for outreach to pregnant women, mothers and children in the communities with the aim to promote safe deliveries as per WHO guidelines and Government policy will be enhanced. In order to deliver quality services, the facilities will be renovated and equipped and the capacity of the existing staff will be strengthened through different training courses in MNCH. In addition professionally trained Lady Health Visitors will be introduced in the BHUs, who will conduct all maternal services including deliveries in the BHU and the communities. The health staff is furthermore responsible to establish and facilitate community support groups and raise communal awareness for the importance of mother and child health care as well as safe deliveries with skilled attendants. Operational research is an integral part of this pilot project. The research validates the progress and improvement of maternal and child health indicators. The results will be used to lobby the scale up of MNCH interventions with the Ministry of Health in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Be a resident of target areas and consent to participate in the study

Exclusion Criteria:

* Do not fulfill the residence and consent criteria

Ages: 1 Day to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15000 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maternal, Neonatal and infant mortality | 24 months
  A 20% reduction in mortality rates is expected

SECONDARY OUTCOMES:
Antenatal Care | 12 months
  A 40% Increase in Antenatal care is expected
Skilled Birth attendance | 12 months
  A 40% increase in Skilled Birth attendance is expected
Essential Neonatal Care | 24 months
  A 40% increase in uptake of Essential Neonatal Care
Child hood Immunization Rates | 24 months
  A 30% increase in child hood immunization rates

CONTACTS AND LOCATIONS:
Overall Officials: Sajid Soofi, FCPS, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: No